CLINICAL TRIAL: NCT05078320
Title: Internet-delivered Cognitive-behaviour Therapy for Adolescents With Body Dysmorphic Disorder: A Feasibility Trial
Brief Title: Internet-delivered Cognitive-behaviour Therapy for Adolescents With Body Dysmorphic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lorena Fernández de la Cruz, PhD, Researcher, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01942
Record Dates: First submitted 2021-09-20; First posted 2021-10-14 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Body Dysmorphic Disorders; Dysmorphophobia
Keywords: Body dysmorphic disorder; Dysmorphophobia; Cognitive-behavioral therapy; Internet-delivered treatments; Adolescents; Treatment outcomes
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-delivered cognitive-behaviour therapy for adolescents with body dysmorphic disorder (Experimental): Cognitive-behaviour therapy, Exposure and response prevention (ERP)
  Interventions: Behavioral: Exposure and response prevention (ERP)

INTERVENTIONS:
Behavioral: Exposure and response prevention (ERP) — The treatment is Internet-delivered and therapist-guided, involving both the adolescent and at least one parent. The treatment consists of two separate sets of modules, one for the adolescent and one for the parent, each with separate logins. The ICBT intervention consists of 12 modules, delivered over a maximum of 14 weeks.
  The main goal of treatment is to help the young person to stop avoiding anxiety-provoking situations by undertaking exposure tasks and to stop doing unhelpful repetitive behaviours and rituals, known as response prevention. Every module also contains homework tasks that mainly consists of exposure and response prevention (ERP).
  Parents are also often involved in the patients' rituals and avoidant behaviours (known as family accommodation), which may contribute to maintain the BDD symptoms. Involving parents facilitates modification of these unhelpful patterns.

SUMMARY:
The purpose of this trial is to investigate whether a therapist-guided Internet-delivered cognitive behaviour therapy (ICBT) programme is feasible for adolescents with body dysmorphic disorder (BDD). The aim is to evaluate feasibility and provide preliminary efficacy data.

DETAILED DESCRIPTION:
Rationale for study: BDD is a prevalent and impairing condition that can be effectively treated with cognitive-behaviour therapy (CBT). However, CBT for BDD is a highly specialised treatment and a majority of adolescents do not have access to it. ICBT can be a way to increase the availability of effective psychological treatments. No study to date has evaluated the feasibility of ICBT for adolescent BDD, but the experience in adults with BDD treated with ICBT is encouraging.

Objectives: To investigate whether a therapist-guided Internet-delivered cognitive behaviour therapy (ICBT) programme is feasible for adolescents with body dysmorphic disorder (BDD). Specifically, the aim is to:(a) establish participant retention, ease of recruitment, acceptability, credibility, and satisfaction, (b) evaluate potential adverse events, and (c) provide preliminary efficacy data.

Trial design and methods: Participants will be recruited nationally and will be offered 12 modules of ICBT for BDD, delivered over a period of 14 weeks. Participants will be assessed before, during, and after treatment, and up to 12 months after the end of the treatment. ICBT non-responders, assessed at post-treatment and one-, two-, and three-months after completing treatment, will be offered CBT delivered via video format (at post-treatment and after the 1MFU and the 2MFU) or traditional face-to-face (F2F) CBT at the OCD and Related Disorders Clinic for Children and Adolescents in Stockholm (after the 3MFU).

The primary outcome is feasibility, as measured by examining rates of participant retention, treatment completion and adherence to treatment content, treatment acceptability, treatment credibility, treatment satisfaction and adverse events during the treatment.

Secondary outcomes include improvement in clinician-reported BDD symptoms, as well as improvement in other clinical measures assessing disorder severity, disorder improvement, self-reported BDD symptoms, depressive symptoms, and functional impairment.

Sample: 20 adolescents and their primary caregivers.

Statistical analysis: Retention, acceptability, credibility, and treatment satisfaction. For retention and acceptability, information on ease of recruitment, number of completed modules, and attrition rates will collected and presented in a descriptive manner. Results from a credibility scale will be summarized in group means and standard deviations. Results from a treatment satisfaction scale will be summarized in group means and standard deviation. Potential adverse events: Type and impact of all potential adverse events will be measured with a specific scale and presented descriptively. Preliminary efficacy: Clinical measures of treatment outcomes will be measured via clinician-reported and self- and parent-reported measures and analysed through linear mixed models to detect within group change over time. Within-group effect sizes will be estimated with Cohen's d. Treatment response: The proportion of treatment responders will be calculated. Treatment response will be defined as a ≥30% reduction on the BDD-YBOCS-A, respective to the baseline score. Further, the investigators will also calculate how many participants are on full or partial symptom remission, defined as a score ⩽16 on the BDD-YBOCS-A.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 to 17 years, confirmed by the caregiver and subsequently by the patient record system Take Care.
2. A diagnosis of BDD, based on the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), confirmed by the assessor at the pre-treatment assessment.
3. A total BDD severity score on the BDD-YBOCS-A ≥24. confirmed by the clinician-reported BDD-YBOCS-A performed at the pre-treatment assessment.
4. A minimum of one available caregiver (parent) to support the child/adolescent throughout the treatment. Confirmed by the caregiver at the telephone screening or/and pre-treatment assessment.
5. Regular access to a desktop or laptop computer connected to the Internet, with the ability to receive e-mails, as well as a mobile phone to receive SMS (one of each per family is enough). Confirmed by the caregiver at the telephone screening or/and pre-treatment assessment.

Exclusion Criteria:

1. Previous CBT for BDD for a minimum of eight sessions with a qualified therapist within the 12 months prior to assessment. Confirmed by the caregiver at the telephone screening and/or pre-treatment assessment.
2. Simultaneous psychological treatment for BDD, confirmed by the caregiver at the telephone screening and/or pre-treatment assessment.
3. Initiation, adjustment or change of any selective serotonin reuptake inhibitors (SSRI) within the six weeks prior to the pre-treatment assessment. Confirmed by the caregiver at the telephone screening and/or pre-treatment assessment.
4. A diagnosis of organic brain disorder, intellectual disability or a psychiatric disorder (such as psychosis, bipolar disorder or eating disorder) that could interfere with the completion of the treatment. Confirmed by the caregiver at the telephone screening and/or pre-treatment assessment, with help of information from the caregiver and the child/adolescent, and the MINI-KID interview.
5. Immediate risk to self or others requiring urgent medical attention, such as current risk of suicide or self-injurious behaviours. Confirmed by the assessor at the telephone screening and/or face-to-face or video conference pre-treatment assessment, with help of information from the caregiver and the child/adolescent, and the suicide questions on the MINI-KID interview.
6. Child and caregiver not able to read and communicate in Swedish. Confirmed by the caregiver or assessor at the telephone screening and/or pre-treatment assessment.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Treatment credibility questionnaire | Mid-treatment (3 weeks post-baseline)
  Questionnaire developed by the research team. Used to assess treatment credibility. Separate versions for the child/adolescent and the parent are used. Range: 0-12, high scores means better outcome.
Treatment satisfaction questionnaire | 3-month follow-up.
  Questionnaire developed by the research team. Used to assess treatment satisfaction. Separate versions for the child/adolescent and the parent are used. Range: 0-36, high scores means better outcome.
internet intervention Patient Adherence Scale (iiPAS) Mid-treatment | Mid-treatment (6 weeks post-baseline)
  Used to assess the child/adolescent's adherence to the internet-delivered treatment. Range: 0-20, high scores means better outcome.
internet intervention Patient Adherence Scale (iiPAS) Post-treatment | Week 14.
  Used to assess the child/adolescent's adherence to the internet-delivered treatment. Range: 0-20, high scores means better outcome.
Negative effects questionnaire - Mid-treatment | Week 6
  Used to assess side effects/adverse events for the child/adolescent. Parent-reported. Range: 0-100, low scores means better outcome.
Negative effects questionnaire - Post-treatment | Week 14
  Used to assess side effects/adverse events for the child/adolescent. Parent-reported. Range: 0-100, low scores means better outcome.
Negative effects questionnaire - 3 months follow-up | 3 months follow-up
  Used to assess side effects/adverse events for the child/adolescent. Parent-reported. Range: 0-100, low scores means better outcome.
Ease of recruitment: Time to recruit | From start of recruitment until 20 participants have been included. Anticipated time frame: 2-3 months
  Time to recruit 20 participants.
Ease of recruitment: Amount of participants accepting participation after screening | From start of recruitment until 20 participants have been included. Anticipated time frame: 2-3 months
  Amount of participants accepting/declining participation after telephone screening
Ease of recruitment: Amount of participants accepting participation after assessment | From start of recruitment until 20 participants have been included. Anticipated time frame: 2-3 months
  Amount of participants accepting/declining participation after initial assessment.
Number of completed chapters in the internet treatment platform | Week 14
  Number of completed chapters is automatically logged in the internet treatment platform. Separate data for children and parents.
Participant retention | Week 14.
  Number of included participants completing treatment.

SECONDARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale Modified for Body Dysmorphic Disorder, Adolescent version (BDD-YBOCS-A) | Baseline; week 14; 1-, 2-, 3-, 6- and 12-month follow-up.
  Used to assess BDD symptom severity. Clinician-rated, semi-structured interview. Range: 0-48, low scores means better outcome.
Clinical Global Impression - Severity (CGI-S) | Baseline; week 14; 3-, 6- and 12-month follow-up.
  Used to provide an overall rating of the BDD severity. Clinician-rated. Range: 1-7, low scores means better outcome.
Clinical Global Impression - Improvement (CGI-I) | Week 14; 3-, 6- and 12-month follow-up.
  Used to assess global improvement. Clinician-rated. Range: 1-7, low scores means better outcome.
Children's Global Assessment Scale (CGAS) | Baseline; week 14; 3-, 6- and 12-month follow-up.
  Used to assess global improvement. Clinician-rated. Range: 1-100, high scores means better outcome.
Appearance Anxiety Index (AAI) | Baseline; week 3, 6, 9, 14; 3-, 6- and 12-month follow-up.
  A self-reported measure that covers cognitions and behaviours typical of BDD. Range: 0-40, low scores means better outcome.
Short Mood and Feeling Questionnaire - child version (SMFQ) + additional suicide item | Baseline; week 3, 6, 9, 14; 3-, 6- and 12-month follow-up.
  Used to assess depressive symptoms and suicidal ideation. Child/adolescent-reported. Range: 0-29, low scores means better outcome.
Short Mood and Feeling Questionnaire - parental version (SMFQ) + additional suicide item | Baseline; week 3, 6, 9, 14; 3-, 6- and 12-month follow-up.
  Used to assess depressive symptoms and suicidal ideation in the adolescent. Parent-reported. Range: 0-29, low scores means better outcome.
The Work and Social Adjustment Scale - Youth Version (WSAS-Y) | Baseline; week 6, 14; 3-, 6- and 12-month follow-up.
  A self-reported instrument assessing functional impairment. Range: 0-40, low scores means better outcome.
The Work and Social Adjustment Scale - Parent Version (WSAS-P) | Baseline; week 6, 14; 3-, 6- and 12-month follow-up.
  A parent-reported instrument assessing functional impairment in the adolescent. Range: 0-40, low scores means better outcome.
CRAFFT (acronym for the key words Car, Relax, Alone, Forget, Friends and Trouble) | Baseline; week 14; 3-, 6- and 12-month follow-up.
  A short self-reported instrument used to identify substance use and substance use disorder. Range: 0-6, low scores means better outcome.
KIDSCREEN-10 | Baseline; week 14; 3-, 6- and 12-month follow-up.
  Used to assess quality of life. Separate versions for the child/adolescent and the parent are used. Range: 10-50, high scores means better outcome.

OTHER OUTCOMES:
Therapist platform time | Week 14
  Therapist platform time is automatically logged in the internet treatment platform. Separate data for children and parents.
Therapist telephone time | Week 14
  Therapist telephone time is manually logged in a spreadsheet throughout the trial. Separate data for children and parents.

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Fernández de la Cruz, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mataix-Cols D, Fernandez de la Cruz L, Isomura K, Anson M, Turner C, Monzani B, Cadman J, Bowyer L, Heyman I, Veale D, Krebs G. A Pilot Randomized Controlled Trial of Cognitive-Behavioral Therapy for Adolescents With Body Dysmorphic Disorder. J Am Acad Child Adolesc Psychiatry. 2015 Nov;54(11):895-904. doi: 10.1016/j.jaac.2015.08.011. Epub 2015 Sep 3. PMID 26506580